CLINICAL TRIAL: NCT03401073
Title: A Double-Blind, Placebo Controlled Trial of Intravenous Immunoglobulin Therapy in Patient With Small Fiber Neuropathy Associated With Autoantibodies to TS-HDS and FGFR3
Brief Title: IVIg for Small Fiber Neuropathy With Autoantibodies TS-HDS and FGFR3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Phoenix Neurological Associates, LTD (Other)
Responsible Party: Principal Investigator, Christopher Gibbons, MD, Associate Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P000592
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Small Fiber Neuropathy; Idiopathic Peripheral Neuropathy
Keywords: small Fiber Neuropathy; Idiopathic Peripheral Neuropathy; IVIg; Gamunex-C
MeSH Terms: conditions — Small Fiber Neuropathy | interventions — Immunoglobulins, Intravenous; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.9% Sodium Chloride (Placebo Comparator): The study will include a total 20 individuals. Subjects will be randomized equally to treatment or placebo. The placebo will consist of 0.9% Sodium Chloride per day over 2 days. Followed by 0.9% Sodium Chloride over 1 day every 3 weeks for a total of 6 treatments. Participants who are randomized to placebo will receive the same volume as they would if they were randomized to IVIG (i.e.: as if receiving IVIG at 2gm/kg) through a peripheral IV line.
  Interventions: Drug: 0.9% Sodium Chloride
- Intravenous Immunoglobulin (Experimental): The study will include a total 20 individuals. Subjects will be randomized equally to treatment or placebo. Treatment will consist of IVIG administered at an initial dose of 2 grams/kg over 2 days followed by 1 gram/kg over 1 day every 3 weeks for a total of 6 treatments
  Interventions: Drug: Intravenous immunoglobulin

INTERVENTIONS:
Drug: Intravenous immunoglobulin — Gamunex-C [immune globulin injection (human) 10% caprylate/chromatography purified] is a sterile solution of human immune globulin protein.
  Other Names: Gamunex-C Liquid
  Arms: Intravenous Immunoglobulin
Drug: 0.9% Sodium Chloride — Sodium Chloride (also known as saline) is a solution of sodium chloride, or salt, and sterile water.
  Other Names: Saline
  Arms: 0.9% Sodium Chloride

SUMMARY:
The objective of this study is to develop a rationale for the selective treatment of small fiber neuropathy with immune globulin (IVIG) in the appropriate patients.

The investigators hypothesize that individuals with auto-antibodies targeting neuronal antigens (TS-HDS and FGFR3) and confirmed evidence of small fiber neuropathy (by skin biopsy analysis of intra-epidermal nerve fiber density) will have an improvement in both nerve fiber density and pain after treatment with immune globulin.

The co-primary endpoints will be a change in neuropathic pain (by VAS pain score) and a change in intra-epidermal nerve fiber density (by punch skin biopsy).

The data gained from this pilot study will establish a rationale, with an appropriate screening test, for the use of immune globulin for the treatment of small fiber neuropathy.

DETAILED DESCRIPTION:
Small fiber neuropathies, and mixed small and large fiber neuropathies, have many potential causes including diabetes, vitamin deficiencies, environmental and toxic exposures, HIV, autoimmune and paraproteinemias.

However, despite this broad differential at least 30% of cases of small fiber neuropathies remain idiopathic. There is therefore a growing interest in the potential for using IVIG in small fiber neuropathy without direct proof that the disorder is caused by immune reactions. We have recently uncovered two novel autoantibodies, TS-HDS and FGFR-3, that are targeted again peripheral neural structure. TS-HDS is a disaccharide component of glycosylation of heparin and heparin sulfate.

Patients with elevated levels of IgM against TS-HDS display clear small fiber loss with IgM deposits around the outside of medium- & larger-sized capillaries with C5b-9 complement deposits. FGFR-3 is a secreted cell surface receptor; genetic defects of FGFR-3 are linked to achrondroplasia and other bony abnormalities.

The antibodies to TS-HDS and FGFR-3 are detected in up to 20% of patients with otherwise idiopathic small fiber neuropathy, but are rare in patients without small fiber neuropathy.

Dr. Levine (a co-investigator on this project) recently presented 3 cases of small fiber associated with elevated levels of auto-antibodies to TS-HDS or FGFR-3 who were treated with IVIG at 2 gm/kg/month for 6 months. He examined skin biopsies for intra-epidermal nerve fiber density and patient self-reported pain scores at baseline and after six months of therapy. All 3 cases showed marked improvement in pain scores. The average reduction in pain was 54%. In addition there was a clear increase in the intra-epidermal nerve fiber density (IENFD) after 6 months of therapy. Pre-treatment IENFD was 1.6, 1.7, and 2.4 at the calf. After 6 months of therapy the IENFD was 8.4, 5.7, 3.3 respectively (these are clinically significant improvement in nerve fiber density.

The investigators believe these anecdotal cases suggest that TS-HDS and FGFR-3 antibodies may be a marker for a group of SFN patients that are immune mediated and may respond to IVIG. (This case series was presented as a poster at the American Academy of Neurology meeting in 2017)

ELIGIBILITY:
Inclusion Criteria:

1. Patient with clinically evident and biopsy proven pure small fiber neuropathy as evidenced by reduced intra-epidermal nerve fiber density seen on skin biopsy using PGP 9.5 as the immunostain.
2. Patients must have a baseline pain score on a VAS scale of Greater or equal to 4/10
3. Patients must have elevated titers of autoantibodies to TS-HDS or FFR3 as measured in Dr Alan Pestronk's lab at Washington University in St Louis.

Exclusion Criteria:

1. Any other known cause for small fiber neuropathy other than the presence of the elevated titers of auto-antibodies. For example patients with diabetes, HIV, Sjogrens, Vitamin deficiency etc.
2. Patients with generalized, severe musculoskeletal conditions other than SFN that prevent a sufficient assessment of the patient by the physician
3. Cardiac insufficiency (New York Heart Association III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease).
4. Severe liver disease (ALAT 3x > normal value).
5. Severe kidney disease (creatinine 1.5x > normal value).
6. Known hepatitis B, hepatitis C or HIV infection.
7. Patients with a history of deep vein thrombosis (DVT) within the last year prior to baseline visit or pulmonary embolism ever; patients with susceptibility to embolism or deep vein thrombosis.
8. Body mass index (BMI) ≥40 kg/m2.
9. Medical conditions whose symptoms and effects could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
10. Known IgA deficiency with antibodies to IgA.
11. History of hypersensitivity, anaphylaxis or severe systemic response to immuno-globulin, blood or plasma derived products, or any component of Gamunex.
12. Known blood hyperviscosity, or other hypercoagulable states.
13. Use of IgG products within six months prior to enrolment.
14. Use of other blood or plasma-derived products within three months prior to enrollment.
15. Patients with a history of drug or alcohol abuse within the past five years prior to enrollment.
16. Patients unable or unwilling to understand or comply with the study protocol
17. Participating in another interventional clinical study with investigational treatment within three months prior to enrollment.
18. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to use an effective birth control method (such as implants, injectable, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner) while on study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gibbons, MD, Principal Investigator — Beth Israel Deaconess Medical Cednter
Locations (1):
- Beth Israel Deaconness Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbons CH. Small fiber neuropathies. Continuum (Minneap Minn). 2014 Oct;20(5 Peripheral Nervous System Disorders):1398-412. doi: 10.1212/01.CON.0000455874.68556.02. PMID 25299289
- [Background] Cortez M, Singleton JR, Smith AG. Glucose intolerance, metabolic syndrome, and neuropathy. Handb Clin Neurol. 2014;126:109-22. doi: 10.1016/B978-0-444-53480-4.00009-6. PMID 25410218
- [Background] Peltier A, Goutman SA, Callaghan BC. Painful diabetic neuropathy. BMJ. 2014 May 6;348:g1799. doi: 10.1136/bmj.g1799. PMID 24803311
- [Background] Kass-Iliyya L, Javed S, Gosal D, Kobylecki C, Marshall A, Petropoulos IN, Ponirakis G, Tavakoli M, Ferdousi M, Chaudhuri KR, Jeziorska M, Malik RA, Silverdale MA. Small fiber neuropathy in Parkinson's disease: A clinical, pathological and corneal confocal microscopy study. Parkinsonism Relat Disord. 2015 Dec;21(12):1454-60. doi: 10.1016/j.parkreldis.2015.10.019. Epub 2015 Nov 3. PMID 26578039
- [Background] Lefaucheur JP, Wahab A, Plante-Bordeneuve V, Sene D, Menard-Lefaucheur I, Rouie D, Tebbal D, Salhi H, Creange A, Zouari H, Ng Wing Tin S. Diagnosis of small fiber neuropathy: A comparative study of five neurophysiological tests. Neurophysiol Clin. 2015 Dec;45(6):445-55. doi: 10.1016/j.neucli.2015.09.012. Epub 2015 Nov 17. PMID 26596193
- [Background] Kafaie J, Al Balushi A, Kim M, Pestronk A. Clinical and Laboratory Profiles of Idiopathic Small Fiber Neuropathy in Children: Case Series. J Clin Neuromuscul Dis. 2017 Sep;19(1):31-37. doi: 10.1097/CND.0000000000000178. PMID 28827487
- [Background] Pestronk A, Schmidt RE, Choksi RM, Sommerville RB, Al-Lozi MT. Clinical and laboratory features of neuropathies with serum IgM binding to TS-HDS. Muscle Nerve. 2012 Jun;45(6):866-72. doi: 10.1002/mus.23256. PMID 22581541
- [Background] Antoine JC, Boutahar N, Lassabliere F, Reynaud E, Ferraud K, Rogemond V, Paul S, Honnorat J, Camdessanche JP. Antifibroblast growth factor receptor 3 antibodies identify a subgroup of patients with sensory neuropathy. J Neurol Neurosurg Psychiatry. 2015 Dec;86(12):1347-55. doi: 10.1136/jnnp-2014-309730. Epub 2015 Jan 27. PMID 25628376
- [Background] Hahn AF, Bolton CF, Zochodne D, Feasby TE. Intravenous immunoglobulin treatment in chronic inflammatory demyelinating polyneuropathy. A double-blind, placebo-controlled, cross-over study. Brain. 1996 Aug;119 ( Pt 4):1067-77. doi: 10.1093/brain/119.4.1067. PMID 8813271
- [Background] Mendell JR, Barohn RJ, Freimer ML, Kissel JT, King W, Nagaraja HN, Rice R, Campbell WW, Donofrio PD, Jackson CE, Lewis RA, Shy M, Simpson DM, Parry GJ, Rivner MH, Thornton CA, Bromberg MB, Tandan R, Harati Y, Giuliani MJ; Working Group on Peripheral Neuropathy. Randomized controlled trial of IVIg in untreated chronic inflammatory demyelinating polyradiculoneuropathy. Neurology. 2001 Feb 27;56(4):445-9. doi: 10.1212/wnl.56.4.445. PMID 11222785
- [Background] Cocito D, Ciaramitaro P, Isoardo G, Barbero P, Migliaretti G, Pipieri A, Proto G, Quadri R, Bergamasco B, Durelli L. Intravenous immunoglobulin as first treatment in diabetics with concomitant distal symmetric axonal polyneuropathy and CIDP. J Neurol. 2002 Jun;249(6):719-22. doi: 10.1007/s00415-002-0698-0. PMID 12111305
- [Background] Eftimov F, Winer JB, Vermeulen M, de Haan R, van Schaik IN. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2013 Dec 30;(12):CD001797. doi: 10.1002/14651858.CD001797.pub3. PMID 24379104
- [Background] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Background] Lauria G, Hsieh ST, Johansson O, Kennedy WR, Leger JM, Mellgren SI, Nolano M, Merkies IS, Polydefkis M, Smith AG, Sommer C, Valls-Sole J; European Federation of Neurological Societies; Peripheral Nerve Society. European Federation of Neurological Societies/Peripheral Nerve Society Guideline on the use of skin biopsy in the diagnosis of small fiber neuropathy. Report of a joint task force of the European Federation of Neurological Societies and the Peripheral Nerve Society. Eur J Neurol. 2010 Jul;17(7):903-12, e44-9. doi: 10.1111/j.1468-1331.2010.03023.x. PMID 20642627
- [Background] Nolano M, Biasiotta A, Lombardi R, Provitera V, Stancanelli A, Caporaso G, Santoro L, Merkies IS, Truini A, Porretta-Serapiglia C, Cazzato D, Dacci P, Vitale DF, Lauria G. Epidermal innervation morphometry by immunofluorescence and bright-field microscopy. J Peripher Nerv Syst. 2015 Dec;20(4):387-91. doi: 10.1111/jns.12146. PMID 26309146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential research subjects were recruited from Beth Israel Deaconess Medical Center (BIDMC) (Boston, MA) and HonorHealth Neurology (Phoenix, AZ). All recruited subjects signed a consent form approved by the Institutional Review Boards of BIDMC and HonorHealth.
Pre-assignment Details: After signing an informed consent, study subjects underwent a detailed history, physical examination, laboratory studies, pain VAS scores, the Short-From 36 question health survey (SF-36), antibody measurement of TS-HDS and FGFR-3 and skin biopsy evaluation of nerve fiber density at the distal leg and proximal thigh using standard methodology.
  If participants did not meet criteria for the study after screening (based on inclusion and exclusion criteria), they were excluded.
Period: Overall Study
Arm/Group | 0.9% Sodium Chloride | Intravenous Immunoglobulin
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% Sodium Chloride | Intravenous Immunoglobulin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (9.4) | 51.5 (7.8) | 51.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Intra-epidermal nerve fiber density [Mean (Standard Deviation); unit: Fibers/mm] | 2.02 (1.49) | 2.47 (1.83) | 2.25 (1.66)
Pain score [Mean (Standard Deviation); unit: units on a scale] | 5.5 (1.2) | 6.9 (1.8) | 6.2 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Nerve Fiber Density Between Visits 1 and 8.
Description: Difference in intra-epidermal nerve fiber density between visits 1 and 8 will be measured.
  Intra-epidermal nerve fiber density is a quantitative measure of the number of nerve fibers per millimeter. The outcome is the number of nerve fibers measured at visit 8 minus the number of nerve fibers measured at visit 1. A positive value indicates that nerve fiber density has increased (a better outcome), a negative value indicates that the nerve fiber density has decreased (a worse outcome).
Time Frame: Visit 1 (time zero) and visit 8 (range of visit time 22-27 weeks after visit 1), thus a total of 22-27 weeks for the study (the range is provided to ensure final follow up is completed despite any conflicts with travel or holidays).
Population: The 17 study completers were analyzed as part of the final results.
Measure: Mean (Standard Deviation); unit: fibers/mm
Arm/Group | 0.9% Sodium Chloride | Intravenous Immunoglobulin
Number analyzed (Participants) | 9 | 8
fibers/mm | 0.5 (0.8) | 0.6 (0.6)

2. Secondary Outcome: The Change in Neuropathic Pain Severity Between Visits 1 and 8.
Description: The visual analog scale (VAS) of pain allows for quantification of neuropathic pain.
  The VAS pain scale depicts a line ranging from 0 (no pain) to 10 (worst possible pain). The scale is ordinal ranging from 0-10.
  The difference in pain between visit 1 and visit 8 (pain measured at visit 8 subtracted from the score at visit 1) is the range. Positive values indicate an increase in pain (worse outcome), negative values indicate an improvement in pain (better outcome).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.9% Sodium Chloride | Intravenous Immunoglobulin
Number analyzed (Participants) | 9 | 8
units on a scale | -1.7 (0.9) | -1.9 (2.6)

3. Secondary Outcome: 2) The Difference in Change Between Quantified Utah Early Neuropathy Examination Scores, Between Treatment and Placebo Groups Between Visits 1 and 8.
Description: The Utah Early Neuropathy Scale (UENS) was developed specifically to detect and quantify early small-fiber sensory neuropathy and to recognize modest changes in sensory severity and distribution.
  The UENS scale ranges from 0 (no neuropathy) to 42 (severe small fiber neuropathy). The outcome measure is the UENS score from Visit 8 minus the UENS score at visit 1. The difference in the two scores indicates the change in neuropathy severity. A positive value indicates that neuropathy has worsened over the course of the study, a negative value indicates that neuropathy has improved over the course of the study.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.9% Sodium Chloride | Intravenous Immunoglobulin
Number analyzed (Participants) | 9 | 8
units on a scale | -3.0 (5.8) | -1.8 (3.9)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events captured at 3 week intervals or by interval phone calls for any acute changes in condition.
Arm/Group | 0.9% Sodium Chloride | Intravenous Immunoglobulin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.9% Sodium Chloride (N=10) | Intravenous Immunoglobulin (N=10)
Infusion reaction (Product Issues) | 9 (25) | 8 (22) — Chills, pain, flushing, tingling, fatigue

LIMITATIONS AND CAVEATS:
This was a small pilot study that was underpowered to detect changes to secondary endpoints.

There was a 15% dropout. Despite several publications that note an association between TS-HDS and FGFR-3 autoantibodies in neuropathy, we do not have evidence for pathogenicity (supported by a non-insignificant number of patients excluded from the study with autoantibodies but without evidence of neuropathy). This too may have limited the potential treatment effect of immune globulin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03401073/Prot_SAP_000.pdf